CLINICAL TRIAL: NCT04938245
Title: Improving Spinal Cord Stimulation With ECAPS
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEUROSURG-2021-29717
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Observed Cohort: Participants with chronic pain scheduled to undergo externalized trial for assessment of spinal cord stimulation will undergo intraoperative stimulation and up to three postoperative visits where already externalized electrodes (used clinically for stimulation) will be used to record and stimulate using evoked complex action potentials (ECAPs) while also measuring other electrophysiological responses.
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Intraoperatively, stimulation at 12 Hz will be performed as the leads are moved into the targeted position. Amplitude will be increased to 15 mA maximum total until a response is seen on any electrode and held for 10 seconds. Stimulation and recording will be performed using the Neuralynx stim/record system.
  Post-operatively, the electrodes will be tested for impedance by the clinical system and then they will be connected to the Neuralynx stim/record system. Electrode stimulation patterns will be applied with increasing amplitude until ECAPs responses are seen on recording electrodes. 42 Hz stimulation will be performed with an amplitude sweep of 0mA-10mA. At each amplitude, stimulation will be applied for 4 seconds followed by 2 seconds of rest. Pulse width will be varied from 30-450 microseconds to test effective amplitude. Bursting stimulation will be applied to detect differences in ECAPs as above.

SUMMARY:
The purpose of this study will be to investigate the optimization of spinal cord stimulation with ECAPs in patients with spinal cord implants.

DETAILED DESCRIPTION:
Spinal cord stimulation (SCS) or electrical stimulation in the epidural space of the spinal canal has been used for more than 50 years to treat chronic pain by modulating the activity of the spinal cord or spinal cord roots. While originally conceived out of gate theory, the precise effects of spinal cord stimulation are still an active area of research. Certainly there are multiple factors contributing to this unchanged responder rate including diagnosis, psychosocial factors, comorbidities, and implementation gaps, but a major technical hurdle remains personalizing therapy to engage in the precise pain circuits for each individual patient in anatomic location and over time. The delivery of spinal cord stimulation varies significantly with changes in position due to the movement of the spinal cord and its associated nerve roots. Existing spinal cord stimulation platforms rely on tonic stimulation with minimal adjustment with movements of the spinal cord or any adjustment due to changing physiology. Tonic stimulation assumes a stationary system that does not account for short or long-term effects of plasticity or movement. However, the effect of stimulation on the circuits of the spinal cord as with all stimulation of the nervous system can be measured through an event-related potential (ERP) synchronized to stimulation pulses, called the evoked compound action potential (ECAP). As an evoked-response, it is clear that ECAPs may provide a more dynamic insight into the underlying electrophysiologic system underlying the anatomic pathways of chronic pain, and some reports have correlated ECAPs to measures of pain relief, which is difficult to disassociate in patients with stable patterns of pain. The spatial variance of ECAP may imply that spinal cord stimulation for the purposes of pain relief is not homologous to features available in the ECAP signal but could be accessible in the variability of ECAP signal. Similarly, very little experimental evidence exists to incorporate the complex role of pain processing and valuation systems into a model of ECAP electrophysiology. Namely, the correlation between top-down control and higher-order (cognitive/mood) circuit interactions with ECAP features and chronic pain. Understanding the electrophysiology of evoked responses in the spinal cord in the competitive market of non-opioid pain relief should be grounded in basic pain phenotype modeling. This proposal represents the first step in that pathway by studying the feasibility of capturing ECAPs during clinical externalization while collecting the necessary data for behavioral modeling for future causal analysis with ECAP features. This protocol establishes the first step towards closed-loop stimulation through open-loop measurement and stimulation during an existing clinical paradigm. This study aims to understand the feasibility of implementing ECAP during the externalization period of a clinical trial while simultaneously providing clinical feedback for optimal settings discovered during testing.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable as determined by the principal investigator
* Scheduled to undergo externalization of spinal cord stimulation
* English-speaking

Exclusion Criteria:

* Scheduled for permanent implantation only without trial
* Have pacemakers or other neurostimulators
* Pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults scheduled to undergo externalization of spinal cord stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Assessed by Enrollment | 2 weeks
  Feasibility will be measured as a number of the number of enrolled participants who complete at least 80% of the planned assessments.

SECONDARY OUTCOMES:
Acceptability Assessed by Survey | 2 weeks
  Acceptability will be measured as the average rating of a five-point qualitative scale ranging from "Excellent" to "Very Poor." Scores range with 1-5 with lower scores indicating greater acceptability.

OTHER OUTCOMES:
Correlation of ECAP peak to peak signals to programming parameters | 2 weeks
Correlation of ECAP signals to pain relief | 2 weeks
Stability and reliability of ECAP sensing | 2 weeks
Reliability of ECAP across various levels intraoperatively | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD, MPH, Principal Investigator — University of Minnesota Medical School Department of Neurosurgery; Alexander Herman, MD, PhD, Principal Investigator — University of Minnesota Medical School Department of Psychiatry; Tay Netoff, PhD, Principal Investigator — University of Minnesota Department of Biomedical Engineering
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
In line with recent requirements of scientific journals, preprocessed and anonymized data will be made available for the research community.
  It will be deposited on the public repository Zenodo (or equivalent) for 5 years.
Time Frame: 5 years

REFERENCES:
- [Derived] Konig S, Ramadan A, Sullivan D, Goel V, Stayner RS, Schultz D, Herman AB, Netoff TI, Darrow DP. Feature extraction and prediction of spinal cord stimulation evoked compound action potentials in humans. J Neural Eng. 2025 Apr 8;22(2). doi: 10.1088/1741-2552/adbfbe. PMID 40073452